CLINICAL TRIAL: NCT01211548
Title: Coronary CT Angiography in Aneurysms Repaired With Open or Endovascular Approach
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 10-573; PVSS1005TM (Other Grant/Funding Number: PVSS)
Record Dates: First submitted 2010-09-09; First posted 2010-09-29 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Complex Aortic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- contrast CTA of the CAP: All patients being considered for a complex aortic surgery and undergoing medically indicated contrast enhanced CT aortic angiography of the chest abdomen and pelvis will be includedRaw data from CT coronary angiography will be available from all patients.
  Interventions: Other: contrast CTA of the CAP

INTERVENTIONS:
Other: contrast CTA of the CAP — CT coronary angiography results will be reported for all patients by adjudicators blinded to their inclusion in the study.

SUMMARY:
This proposal is for the pilot study that will inform the conduct of a larger prospective randomized controlled trial to guide perioperative work up and the cost/utility of CTCA (high definition CT coronary angiography.)

DETAILED DESCRIPTION:
This proposal is for a pilot study that will inform the conduct of a prospective, blinded randomized controlled trial designed to determine the cost effectiveness of an algorithm for pre operative cardiac risk stratification that uses coronary CT angiography. In addition perioperative and long-term cardiac event rate will be recorded to determine if there is any difference in these rates between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* patients being considered for a complex aortic surgery and undergoing medically indicated contrast enhanced CT aortic angiography of the chest abdomen and pelvis

Exclusion Criteria:

* Patients with contraindications to undergoing CT coronary angiography
* coronary revascularization within the last six months
* renal dysfunction in whom the treating physician has decided a contrast enhanced CT scan is not warranted as part of the routine clinical work up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients being considered for a complex aortic surgery and undergoing medically indicated contrast enhanced CT aortic angiography of the chest abdomen and pelvis will be includedRaw data from CT coronary angiography will be available from all patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome for the pilot study will be to assess feasibility of processes as set out in the specific aims. | 6 months

IPD SHARING:
Plan to Share IPD: No